CLINICAL TRIAL: NCT02519036
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Doses of Intrathecally Administered ISIS 443139 in Patients With Early Manifest Huntington's Disease
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ISIS 443139 in Participants With Early Manifest Huntington's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 443139-CS1; 2015-000381-66 (EudraCT Number)
Record Dates: First submitted 2015-08-01; First posted 2015-08-10 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Huntington's Disease
Keywords: Huntington's Disease; HTTRx; Early Manifest Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — HTT(RX)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: Yes

ARMS (6):
- ISIS 443139 10 mg (Experimental): Participants received ISIS 443139, 10 milligrams (mg), by intrathecal injection, on Study Days 1, 29, 57, and 85.
  Interventions: Drug: ISIS 443139 10 mg
- ISIS 443139 30 mg (Experimental): Participants received ISIS 443139, 30 mg, by intrathecal injection, on Study Days 1, 29, 57, and 85.
  Interventions: Drug: ISIS 443139 30 mg
- ISIS 443139 60 mg (Experimental): Participants received ISIS 443139, 60 mg, by intrathecal injection, on Study Days 1, 29, 57, and 85.
  Interventions: Drug: ISIS 443139 60 mg
- ISIS 443139 90 mg (Experimental): Participants received ISIS 443139, 90 mg, by intrathecal injection, on Study Days 1, 29, 57, and 85.
  Interventions: Drug: ISIS 443139 90 mg
- ISIS 443139 120 mg (Experimental): Participants received ISIS 443139, 120 mg, by intrathecal injection, on Study Days 1, 29, 57, and 85.
  Interventions: Drug: ISIS 443139 120 mg
- Placebo (Placebo Comparator): Participants received placebo, by intrathecal injection, on Study Days 1, 29, 57, and 85.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ISIS 443139 10 mg — ISIS 443139, 10 mg, was administered by intrathecal injection, on Study Days 1, 29, 57, and 85.
  Other Names: IONIS HTTRx
  Arms: ISIS 443139 10 mg
Drug: ISIS 443139 30 mg — ISIS 443139, 30 mg, was administered by intrathecal injection, on Study Days 1, 29, 57, and 85.
  Other Names: IONIS HTTRx
  Arms: ISIS 443139 30 mg
Drug: ISIS 443139 60 mg — ISIS 443139, 60 mg, was administered by intrathecal injection, on Study Days 1, 29, 57, and 85.
  Other Names: IONIS HTTRx
  Arms: ISIS 443139 60 mg
Drug: ISIS 443139 90 mg — ISIS 443139, 90 mg, was administered by intrathecal injection, on Study Days 1, 29, 57, and 85.
  Other Names: IONIS HTTRx
  Arms: ISIS 443139 90 mg
Drug: ISIS 443139 120 mg — ISIS 443139, 120 mg, was administered by intrathecal injection, on Study Days 1, 29, 57, and 85.
  Other Names: IONIS HTTRx
  Arms: ISIS 443139 120 mg
Other: Placebo — Placebo was administered by intrathecal injection, on Study Days 1, 29, 57, and 85.
  Arms: Placebo

SUMMARY:
This study tested the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple ascending doses of ISIS 443139 administered intrathecally to adult participants with early manifest Huntington's Disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with early manifest Huntington's disease
* Male or female, aged 25 to 65 years, inclusive, at the time of informed consent
* Able and willing to meet all study requirements, including travel to Study Center and participation in all procedures and measurements at study visits
* Have a trial partner who is reliable, competent and at least 18 years of age, is willing to accompany the participant to select trial visits and to be available to the Study Center by phone if needed
* Able to tolerate MRI scans, blood draws and lumbar punctures
* Reside within 4 hours travel of the Study Center

Key Exclusion Criteria:

* Clinically significant medical condition, such as severe chorea, active suicidal ideation or any other conditions which would make the participant unsuitable for inclusion or could interfere with the participant participating in or completing the study
* Recent treatment with another investigational drug, biological agent, or device
* Prior treatment with an antisense oligonucleotide [including small interfering ribonucleic acid (siRNA)]
* Any history of gene therapy or cell transplantation or any other experimental brain surgery
* Presence of an implanted shunt for the drainage of cerebrospinal fluid (CSF) or an implanted central nervous system (CNS) catheter
* History of post-lumbar-puncture headache of moderate or severe intensity and/or blood patch
* Malignancy within 5 years of Screening, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated
* Hospitalization for any major medical or surgical procedure involving general anesthesia within 12 weeks of Screening or planned during the study

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-08-06 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- University of British Columbia, Vancouver, British Columbia, Canada
- Germany (3):
  - Charite University Berlin, Berlin
  - Ruhr-University of Bochum, Bochum
  - Ulm University Hospital, Ulm
- United Kingdom (5):
  - University Hospitals Birmingham, Birmingham
  - Cambridge University Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - University College London, London
  - University of Manchester, St. Mary's Hospital, Manchester

REFERENCES:
- [Derived] Rodrigues FB, Ferreira JJ, Wild EJ. Huntington's Disease Clinical Trials Corner: June 2019. J Huntingtons Dis. 2019;8(3):363-371. doi: 10.3233/JHD-199003. PMID 31381524
- [Derived] Tabrizi SJ, Leavitt BR, Landwehrmeyer GB, Wild EJ, Saft C, Barker RA, Blair NF, Craufurd D, Priller J, Rickards H, Rosser A, Kordasiewicz HB, Czech C, Swayze EE, Norris DA, Baumann T, Gerlach I, Schobel SA, Paz E, Smith AV, Bennett CF, Lane RM; Phase 1-2a IONIS-HTTRx Study Site Teams. Targeting Huntingtin Expression in Patients with Huntington's Disease. N Engl J Med. 2019 Jun 13;380(24):2307-2316. doi: 10.1056/NEJMoa1900907. Epub 2019 May 6. PMID 31059641
- [Derived] Rodrigues FB, Wild EJ. Huntington's Disease Clinical Trials Corner: February 2018. J Huntingtons Dis. 2018;7(1):89-98. doi: 10.3233/JHD-189001. PMID 29480210
- See also: Ionis Pharmaceuticals, Inc. home page — http://www.ionispharma.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 46 participants were enrolled in the United Kingdom, Canada and Germany.
Groups:
- Placebo: Participants received placebo, by intrathecal injection, at 4 week intervals over the course of a 13 week treatment period.
- ISIS 443139 10 mg: Participants received ISIS 443139, 10 milligrams (mg), by intrathecal injection, at 4 week intervals over the course of a 13 week treatment period.
- ISIS 443139 30 mg: Participants received ISIS 443139, 30 mg, by intrathecal injection, at 4 week intervals over the course of a 13 week treatment period.
- ISIS 443139 60 mg: Participants received ISIS 443139, 60 mg, by intrathecal injection, at 4 week intervals over the course of a 13 week treatment period.
- ISIS 443139 90 mg: Participants received ISIS 443139, 90 mg, by intrathecal injection, at 4 week intervals over the course of a 13 week treatment period.
- ISIS 443139 120 mg: Participants received ISIS 443139, 120 mg, by intrathecal injection, at 4 week intervals over the course of a 13 week treatment period.
Period: Overall Study
Arm/Group | Placebo | ISIS 443139 10 mg | ISIS 443139 30 mg | ISIS 443139 60 mg | ISIS 443139 90 mg | ISIS 443139 120 mg
Started | 12 | 3 | 6 | 6 | 9 | 10
Completed | 12 | 3 | 6 | 6 | 9 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who were randomized and received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ISIS 443139 10 mg | ISIS 443139 30 mg | ISIS 443139 60 mg | ISIS 443139 90 mg | ISIS 443139 120 mg | Total
Number analyzed (Participants) | 12 | 3 | 6 | 6 | 9 | 10 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (10) | 44 (17) | 53 (7) | 43 (11) | 46 (10) | 45 (10) | 47 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 1 | 3 | 3 | 6 | 18
  Male | 8 | 2 | 5 | 3 | 6 | 4 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 3 | 5 | 6 | 9 | 9 | 43
  Black | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Other Race | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 12 | 3 | 6 | 6 | 9 | 10 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events (TEAEs)
Description: An adverse event (AE) was any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE was considered related to the investigational drug product. An AE was to be regarded as a TEAE if it was present prior to receiving the first dose of Study Drug and subsequently worsened or was not present prior to receiving the first dose of Study Drug but subsequently appeared.
Time Frame: Up to approximately 28 weeks
Population: Safety set included all participants who were randomized and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ISIS 443139 10 mg | ISIS 443139 30 mg | ISIS 443139 60 mg | ISIS 443139 90 mg | ISIS 443139 120 mg
Number analyzed (Participants) | 12 | 3 | 6 | 6 | 9 | 10
Participants | 12 | 3 | 6 | 6 | 9 | 9

2. Secondary Outcome: Observed Cerebrospinal Fluid (CSF) Concentration for ISIS 443139
Time Frame: Days 1, 29, 57, 85, and 113 or 141
Population: Pharmacokinetic (PK) population included all participants who were randomized to ISIS 443139, received at least one dose and had sufficient sampling to permit PK evaluation.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | ISIS 443139 10 mg | ISIS 443139 30 mg | ISIS 443139 60 mg | ISIS 443139 90 mg | ISIS 443139 120 mg
Number analyzed (Participants) | 3 | 6 | 6 | 9 | 10
nanograms per milliliter (ng/mL)
  Day 1 | NA (NA) — 'NA' signifies that the values were below the lower limit of quantitation. | NA (NA) — 'NA' signifies that the values were below the lower limit of quantitation. | NA (NA) — 'NA' signifies that the values were below the lower limit of quantitation. | NA (NA) — 'NA' signifies that the values were below the lower limit of quantitation. | NA (NA) — 'NA' signifies that the values were below the lower limit of quantitation.
  Day 29 | NA (NA) — 'NA' signifies that the values were below the lower limit of quantitation. | NA (NA) — 'NA' signifies that the values were below the lower limit of quantitation. | 1.77 (1.61) | 1.55 (1.06) | 2.06 (1.01)
  Day 57 | NA (NA) — 'NA' signifies that the values were below the lower limit of quantitation. | 1.69 (0.530) | 2.77 (2.04) | 2.36 (1.34) | 2.40 (1.24)
  Day 85 | NA (NA) — 'NA' signifies that the values were below the lower limit of quantitation. | 1.96 (1.22) | 2.88 (2.54) | 2.05 (1.25) | 2.53 (0.628)
  Day 113: number analyzed (Participants) | 3 | 3 | 3 | 5 | 5
  Day 113 | NA (NA) — 'NA' signifies that the values were below the lower limit of quantitation. | 1.63 (0.250) | 1.84 (1.71) | 2.28 (0.438) | 2.70 (1.20)
  Day 141: number analyzed (Participants) | 0 | 3 | 3 | 4 | 5
  Day 141 |  | NA (NA) — 'NA' signifies that the values were below the lower limit of quantitation. | NA (NA) — 'NA' signifies that the values were below the lower limit of quantitation. | NA (NA) — 'NA' signifies that the values were below the lower limit of quantitation. | NA (NA) — 'NA' signifies that the values were below the lower limit of quantitation.

3. Other Pre Specified Outcome: Maximum Plasma Concentration (Cmax) for ISIS 443139
Time Frame: Days 1 and 85
Population: PK population included all participants who were randomized to ISIS 443139, received at least one dose and had sufficient sampling to permit PK evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ISIS 443139 10 mg | ISIS 443139 30 mg | ISIS 443139 60 mg | ISIS 443139 90 mg | ISIS 443139 120 mg
Number analyzed (Participants) | 3 | 6 | 6 | 9 | 10
ng/mL
  Day 1 | 74.0 (24.3) | 203 (81.9) | 500 (39.0) | 600 (94.9) | 717 (69.2)
  Day 85 | 124 (73.6) | 179 (55.1) | 396 (77.2) | 439 (86.0) | 731 (90.6)

4. Other Pre Specified Outcome: Time to Maximum Plasma Concentration (Tmax) for ISIS 443139
Time Frame: Days 1 and 85
Population: as for outcome 3
Measure: Median (Full Range); unit: hour (h)
Arm/Group | ISIS 443139 10 mg | ISIS 443139 30 mg | ISIS 443139 60 mg | ISIS 443139 90 mg | ISIS 443139 120 mg
Number analyzed (Participants) | 3 | 6 | 6 | 9 | 10
hour (h)
  Day 1 | 3.03 [2.05 to 5.95] | 3.03 [2.00 to 4.00] | 1.99 [0.533 to 3.08] | 3.05 [2.00 to 8.02] | 4.00 [2.00 to 23.8]
  Day 85 | 2.02 [0.717 to 3.02] | 2.03 [0.550 to 3.07] | 2.02 [1.00 to 4.02] | 3.02 [0.600 to 5.02] | 4.03 [2.00 to 23.9]

5. Other Pre Specified Outcome: Change From Baseline in CSF Mutant Huntingtin (fM) Protein Concentration
Description: Baseline was defined as the last non-missing measure prior to the first dose.
Time Frame: Baseline to Final Assessment (Day 85 or 113)
Population: Per protocol set included all participants who were randomized and received all doses of the protocol-specified study drug.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | ISIS 443139 10 mg | ISIS 443139 30 mg | ISIS 443139 60 mg | ISIS 443139 90 mg | ISIS 443139 120 mg
Number analyzed (Participants) | 12 | 3 | 6 | 6 | 9 | 10
ng/mL
  Baseline | 109.13 (42.57) | 143.65 (49.74) | 119.83 (45.27) | 116.70 (30.46) | 104.99 (65.01) | 95.87 (35.11)
  Change from Baseline | 4.08 (28.47) | -31.28 (25.71) | -31.98 (24.96) | -30.83 (17.17) | -45.76 (27.65) | -38.41 (21.59)

6. Other Pre Specified Outcome: Change From Baseline in CSF Neurofilament Light Chain Concentration
Description: Baseline was defined as the last non-missing measure prior to the first dose.
Time Frame: Baseline to Final Assessment (Day 85 or 113)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nanograms per liter (ng/L)
Arm/Group | Placebo | ISIS 443139 10 mg | ISIS 443139 30 mg | ISIS 443139 60 mg | ISIS 443139 90 mg | ISIS 443139 120 mg
Number analyzed (Participants) | 12 | 3 | 6 | 6 | 9 | 10
nanograms per liter (ng/L)
  Baseline | 2774 (767) | 2697 (1909) | 2548 (916) | 2280 (976) | 2328 (951) | 2551 (872)
  Change from Baseline | 324 (371) | 77 (223) | 202 (493) | 274 (301) | 1161 (2980) | 628 (1128)

7. Other Pre Specified Outcome: Ventricular Volume as Assessed by Structural Magnetic Resonance Imaging (MRI)
Time Frame: Screening, Days 113, and 197
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | ISIS 443139 10 mg | ISIS 443139 30 mg | ISIS 443139 60 mg | ISIS 443139 90 mg | ISIS 443139 120 mg
Number analyzed (Participants) | 12 | 3 | 6 | 6 | 9 | 10
mL
  Screening | 35.58 (19.02) | 17.88 (12.20) | 33.02 (17.46) | 31.90 (13.21) | 39.33 (23.52) | 27.53 (19.31)
  Day 113 | 36.11 (19.37) | 18.66 (12.84) | 33.56 (17.87) | 32.04 (14.26) | 42.24 (25.80) | 30.36 (21.80)
  Day 197 | 36.46 (18.97) | 19.69 (13.03) | 34.82 (18.16) | 34.57 (14.82) | 44.43 (27.37) | 33.02 (24.61)

8. Other Pre Specified Outcome: Huntington's Disease (HD) Cognitive Assessment Battery Composite Score
Description: The HD Cognitive Battery was developed as a means of measuring cognitive dysfunction in late premanifest and early manifest HD patients. The 6 tests that comprise the battery were selected based on test sensitivity, practice effects, reliability, domain coverage, feasibility for use in clinical trials, and tolerability. A composite cognitive score was calculated by the average z-score of the 6 individual tests. A positive change from baseline indicated improvement in cognitive function; a negative change indicated worsening. Baseline was defined as the last non-missing measure prior to the first dose.
Time Frame: Baseline to Days 84, 141, and 197
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | ISIS 443139 10 mg | ISIS 443139 30 mg | ISIS 443139 60 mg | ISIS 443139 90 mg | ISIS 443139 120 mg
Number analyzed (Participants) | 12 | 3 | 6 | 6 | 9 | 10
score on a scale
  Baseline | -0.0860 (0.2941) | 0.2979 (0.5157) | 0.0839 (0.5108) | -0.0404 (0.3976) | -0.1483 (0.3284) | 0.1212 (0.3877)
  Change at Day 84 | -0.0403 (0.2261) | 0.1314 (0.3670) | -0.0430 (0.3585) | -0.0338 (0.2756) | 0.1297 (0.2560) | -0.0920 (0.1668)
  Change at Day 141: number analyzed (Participants) | 12 | 3 | 6 | 6 | 9 | 8
  Change at Day 141 | 0.0432 (0.1829) | 0.4441 (0.8487) | -0.1065 (0.2112) | -0.1792 (0.2298) | 0.2194 (0.2224) | -0.0547 (0.2136)
  Change at Day 197: number analyzed (Participants) | 11 | 3 | 6 | 5 | 7 | 10
  Change at Day 197 | -0.0778 (0.2881) | 0.4202 (1.0482) | -0.0469 (0.3151) | -0.1633 (0.1170) | 0.0827 (0.2897) | -0.1387 (0.2717)

ADVERSE EVENTS:
Time Frame: Up to approximately 28 weeks
Description: Safety set included all participants who were randomized and received at least one dose of study drug.
Arm/Group | Placebo | ISIS 443139 10 mg | ISIS 443139 30 mg | ISIS 443139 60 mg | ISIS 443139 90 mg | ISIS 443139 120 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/3 | 0/6 | 0/6 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/3 | 0/6 | 0/6 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 12/12 | 3/3 | 6/6 | 6/6 | 9/9 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | ISIS 443139 10 mg (N=3) | ISIS 443139 30 mg (N=6) | ISIS 443139 60 mg (N=6) | ISIS 443139 90 mg (N=9) | ISIS 443139 120 mg (N=10)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | ISIS 443139 10 mg (N=3) | ISIS 443139 30 mg (N=6) | ISIS 443139 60 mg (N=6) | ISIS 443139 90 mg (N=9) | ISIS 443139 120 mg (N=10)
Procedural pain (Injury, poisoning and procedural complications) | 6 | 1 | 1 | 3 | 6 | 8
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 4 | 1 | 2 | 1 | 3 | 5
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 1 | 2 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Tooth injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 1 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 3 | 1 | 0
Rhinitis (Infections and infestations) | 2 | 0 | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 6 | 0 | 1 | 1 | 1 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleocytosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 1 | 2 — General disorders and administration site conditions
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 — General disorders and administration site conditions
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 — General disorders and administration site conditions
Discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 — General disorders and administration site conditions
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 — General disorders and administration site conditions
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 — General disorders and administration site conditions
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Thyroxine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Urine analysis abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 2 | 1 | 0 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
There are no limitations or caveats for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT02519036/Prot_SAP_000.pdf